CLINICAL TRIAL: NCT01317394
Title: Retrospective Study and Analysis of Micafungin for Non-albican Candidemia: Efficacy, Risk Factor and Clinical Manifestation
Brief Title: Study and Analysis of Micafungin for Non-albican Candidemia: Efficacy, Risk Factor and Clinical Manifestation
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Wen-Sen Lee, Department of Infectious Disease, WanFang Hospital
Other Study IDs: 99078
Record Dates: First submitted 2011-03-15; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Non-albicans Candidemia
Keywords: non-albicans candidemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a retrospective research in order to compare and analysis the risk factor, clinical manifestation and efficacy of albicans candidemia by pulling medical records. We hope that this retrospective research will let us understand the method of treatment and prevention of albicans candidemia in order to improve the quality of healthcare.

ELIGIBILITY:
Inclusion Criteria:

* above 20 years old
* hospital patients
* albicans candidemia patients

Exclusion Criteria:

* pregnant patients or patients under 16 years old
* liver cirrhosis and Child C

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-albicans candidemia patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-12; Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Sen Lee, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan